CLINICAL TRIAL: NCT06830928
Title: Validity and Reliability of the PhysioMaster Application in Measuring Wrist Range of Motion (ROM) Among Healthy Adults
Acronym: PhysioMaster
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Abd el fattah Ali, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Other Study IDs: P.T.REC/012/005540
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: PhysioMaster Application in Measuring Wrist Range of Motion (ROM)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Universal Goniometer (UG) is a well-established tool for measuring joint range of motion (ROM). However, it presents limitations, including dependence on examiner skill, which can introduce error. With advances in digital technology, smartphone-based applications, such as PhysioMaster, now offer an alternative approach that potentially reduces human error and increases measurement precision

DETAILED DESCRIPTION:
Measuring Wrist ROM Using the electronic Goniometer

The following protocol will be implemented to measure wrist ROM for the enrolled female participants:

Wrist Flexion-Extension Testing Position: Elbow flexed at 90 degrees, with the wrist positioned over the edge of a table and the forearm in full pronation.

Goniometer Axis: Lateral placement over the triquetrum. Stationary Arm: Aligned with the lateral midline of the ulna, directed toward the olecranon process.

Moving Arm: Aligned with the lateral midline of the 5th metacarpal. Wrist Radial-Ulnar Deviation Testing Position: Elbow flexed at 90 degrees, wrist positioned over the edge of a table with the forearm in full pronation.

Goniometer Axis: Positioned over the dorsal capitate. Stationary Arm: Aligned with the dorsal midline of the forearm. Moving Arm: Positioned parallel to the longitudinal axis of the third metacarpal (Surangsrirat et al., 2022).

Measurement using the smartphone inclinometer-based application For measurements using the smartphone inclinometer application, the smartphone was placed on the participant's wrist, with elbows and upper arms positioned against a wall and flat along their torsos for each movement. This standardized setup ensured consistent smartphone positioning across all ROM measurements .

ELIGIBILITY:
Inclusion Criteria:

- A sample of 30 female participants, aged 19 to 50 years, was selected for this study. Inclusion criteria required participants to be within this age range

Exclusion Criteria:

* any wrist pain, rheumatoid conditions, trauma, prior hand surgeries, deformities in either hand, or pregnancy

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A sample of 30 female participants, aged 19 to 50 years, was selected for this study. Inclusion criteria required participants to be within this age range and free from any wrist pain, rheumatoid conditions, trauma, prior hand surgeries, deformities in either hand, or pregnancy
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-08 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
wrist rane of motion | 4 weeks
  This study employed the digital Goniometer to measure wrist Range of Motion (ROM) in terms of extension, flexion, radial deviation, and ulnar deviation. Additionally, a smartphone inclinometer-based application, PhysioMaster, was used as a comparative tool, compatible with both Android and iOS systems